CLINICAL TRIAL: NCT06060314
Title: Comparison of Efficacy Between Conservative Versus Operative Management of Carpel Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Muhammad Adnan Afsar, Major Doctor, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Combined Military Hospital Ab
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Splints

STUDY DESIGN:
Intervention Model Description: This was a randomized control trial. To ensure randomization, the lottery method was used to allocate the patients to study groups. Patients in Group A were treated conservatively i.e Splinting in neutral position of wrist for 6 wks min at night and during the day as preferred while patients in Group B were managed through surgical intervention i.e open carpal tunnel release (OCTR). Patients were assessed during a follow up visit at 3rd month measured using functional status scale of the Boston questionnaire (BQ).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients presented with symptoms of numbness at night, pain, or tingling sensation in the fingers particularly at night diagnosed by consultant orthopedic surgeon on physical examination. To ensure randomization, the lottery method was used to allocate the patients to study groups. Patients in Group A were treated conservatively i.e Splinting in neutral position of wrist for 6 wks min at night and during the day as preferred while patients in Group B were managed through surgical intervention i.e open carpal tunnel release (OCTR). Patients were assessed during a follow up visit at 3rd month measured using functional status by consultant orthopedic surgeon. Data was recorded by the principle investigator under the supervision of consultant orthopedic surgeon.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients (Other): Patients presented with symptoms of numbness at night, pain, or tingling sensation in the fingers particularly at night diagnosed by a consultant orthopedic surgeon on physical examination.
  Interventions: Procedure: Conservative Approach; Procedure: Surgical Approach
- Principle Investigator (Other): The principal investigator will carry out the whole study.
  Interventions: Procedure: Conservative Approach; Procedure: Surgical Approach
- Consultant Orthopedic Surgeon (Other): Consultant Orthopedic Surgeon will be outcome assessor.
  Interventions: Procedure: Conservative Approach; Procedure: Surgical Approach

INTERVENTIONS:
Procedure: Conservative Approach — Patients in Group A were treated conservatively i.e Splinting in neutral position of wrist for 6 wks min at night and during the day as preferred
  Other Names: Splinting
Procedure: Surgical Approach — Patients in Group B were managed through surgical intervention i.e open carpal tunnel release (OCTR)
  Other Names: open carpal tunnel release (OCTR)

SUMMARY:
Patients presented with symptoms of numbness at night, pain, or tingling sensation in the fingers particularly at night diagnosed by consultant orthopedic surgeon on physical examination. Patients in Group A were treated conservatively i.e splinting in neutral position of wrist for 6 wks min at night and during the day as preferred while patients in Group B were managed through surgical intervention i.e open carpal tunnel release (OCTR). Patients were assessed during a follow up visit at 3rd month measured using functional status scale of the Boston questionnaire (BQ). Efficacy was determined in terms of functional improvement from the baseline.

DETAILED DESCRIPTION:
This randomized controlled trial was conducted at the Department of Orthopedic Surgery, CMH Abbottabad, from 3 March 2022 to 3 September 2022. Ethical approval (file no: CMH-ADT-73-Ortho-23) was sought from the Ethical Committee.

The sample size was calculated by WHO Sample Size calculator with 90% 10 efficacy of surgical treatment and 59.1% 11 efficacy of conservative treatment, with 80% power of test and 5% significance level. Nonprobability consecutive sampling technique was used to gather the sample for this trial.

Inclusion Criteria: Patients of either gender, aged between 18 to 60 years presented with symptoms of numbness at night, pain, or tingling sensation in the fingers particularly at night diagnosed for Carpal tunnel syndrome (CTS) by consultant orthopedic surgeon on physical examination were included in the study.

Exclusion Criteria: Patients already under treatment for carpal tunnel syndrome (CTS) were excluded.

Written informed consent was also taken from all the study participants after a complete description. Carpal tunnel syndrome (CTS) was diagnosed by consultant orthopedic surgeon on physical examination having symptoms of numbness at night, pain, or tingling sensation in the fingers particularly at night. To ensure randomization, the lottery method was used to allocate the patients to study groups. Patients in Group A were treated conservatively i.e Splinting in neutral position of wrist for 6 wks min at night and during the day as preferred while patients in Group B were managed through surgical intervention i.e open carpal tunnel release (OCTR). Patients were assessed during a follow up visit at 3rd month measured using functional status scale of the Boston questionnaire (BQ). The Functional Status Scale (FSS) from the Boston Carpal Tunnel Questionnaire is an 8-item questionnaire originally developed by Levine et al. [10] to assess functional abilities in patients with CTS. Each item of the FSS is rated on a scale from "1" "no difficulty" to "5" "unable." The overall score for the FSS was calculated as the mean of the completed items, and ranges from 1 to 5. Higher scores indicated greater disability. Efficacy was determined in terms of functional improvement from the baseline. An improvement of '2' points from the baseline was termed efficacious.

ELIGIBILITY:
Inclusion Criteria:

Patients of either gender, aged between 18 to 60 years presented with symptoms of numbness at night, pain, or tingling sensation in the fingers particularly at night diagnosed for Carpal tunnel syndrome (CTS) by a consultant orthopedic surgeon on physical examination were included in the study.

Exclusion Criteria:

Patients already under treatment for carpal tunnel syndrome (CTS) were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-09-03 (Actual)

PRIMARY OUTCOMES:
Efficacy in terms of Functional Status Scale Score (FSS Score) | 3 months
  Efficacy was determined in terms of functional improvement from the baseline as per Functional Status Scale Score

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ad Afsar, Principal Investigator — Combined Military Hospital Abbottabad
Locations (1):
- Combined Military Hospital Abbottabad, Abbottabad, Khyber Pukhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
I am not going to share it with other researchers.